CLINICAL TRIAL: NCT07051096
Title: Responsive Nature-Driven Imagery to Reduce Delirium After Cardiac Surgery: A Pilot Randomized Controlled Trial
Brief Title: Responsive Nature-Driven Imagery to Reduce Delirium After Cardiac Surgery
Acronym: RESPITE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Anesthesiologists' Society (Other)
Responsible Party: Principal Investigator, Alana Flexman, Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H24-03693
Record Dates: First submitted 2025-06-19; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Delirium - Postoperative; Agitation; Anxiety; Cardiac Surgery Recovery
Keywords: Randomized trial; Delirium; Cardiac surgery; MindfulGarden
MeSH Terms: conditions — Emergence Delirium; Psychomotor Agitation; Anxiety Disorders; Delirium

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to either the intervention (MindfulGarden) or standard of care. Due to the nature of the intervention, blinding is not possible. In the intervention group, MindfulGarden will be available to participants for the first 7 days after surgery or until discharge, whichever comes first. In both groups, participants will receive standard post-surgical care and routine non-pharmacological delirium reduction measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Receives the MindfulGarden intervention in addition to routine post-operative management and standard delirium reduction measures.
  Interventions: Device: A novel device developed providing nature-driven responsive imagery that responds to the patient's physiological to distract, engage, and de-escalate behaviours of delirium.
- Control Group (Active Comparator): Participants will receive standard care, which includes routine post-operative care pathways for cardiac surgery, and standard delirium reduction measures.
  Interventions: Procedure: Routine post-operative management and standard delirium reduction measures.

INTERVENTIONS:
Device: A novel device developed providing nature-driven responsive imagery that responds to the patient's physiological to distract, engage, and de-escalate behaviours of delirium. — This device will be provided on top of routine post-operative management and standard delirium reduction measures. It has proven effective in a previous clinical trial by reducing agitation and unscheduled medications. It displays nature-driven responsive imagery through an available mobile screen/device for the first 7 days after surgery or discharge, whichever comes first. The imagery adapts in real-time to the participant's movement and sound. The device will be placed at the foot of the bed while the patient is awake and may be interrupted at the discretion of the patient, bedside RN or attending physician.
  Other Names: MindfulGarden
  Arms: Intervention Group
Procedure: Routine post-operative management and standard delirium reduction measures. — Examples of routine post-operative care are sleep optimization, avoidance of delirium-promoting medications, orientation, and mobilization.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to learn if a novel device (MindfulGarden) is beneficial in a population of patients undergoing cardiac surgery. The main questions it aims to answer are:

Is a novel device (MindfulGarden) that uses responsive nature-driven imagery feasible in patients undergoing cardiac surgery? Will use of this device reduce the use of psychotropic medications, improve recovery experience, and improve delirium?

Participants will receive routine post-operative management and standard delirium reduction measures. They will be randomized into two groups where one receives the novel device (MindfulGarden) and the other does not.

DETAILED DESCRIPTION:
Hypotheses:

This study will explore: (1) the feasibility of using Mindful Garden-a novel, nature-based digital therapeutic device offering responsive imagery and sound with biofeedback-in patients undergoing cardiac surgery; and (2) whether its use reduces psychotropic medication use, agitation, anxiety, and both the incidence and duration of postoperative delirium.

Rationale:

Delirium is a frequent, serious complication after cardiac surgery, leading to prolonged hospital stays, increased costs, and higher mortality rates. Although medications are often used to manage delirium-related behavior, they can lead to over-sedation and do not reliably prevent or treat delirium. There is an urgent need for safe, effective, non-pharmacological interventions in high-risk groups. Mindful Garden offers a screen-based display of dynamic nature scenes with interactive elements that respond to physiological cues. In prior ICU settings, brief exposure to Mindful Garden reduced agitation and the need for unscheduled medications. However, its effectiveness in preventing or managing delirium specifically in cardiac surgical patients remains unexplored.

Objectives:

The primary goals are to evaluate the feasibility of implementing Mindful Garden (in terms of recruitment, adherence, data completeness), its usage patterns, and patient satisfaction. Secondary aims include assessing the device's impact on delirium incidence and severity, need for psychotropic medications, agitation levels, anxiety, postoperative recovery, and length of hospital stay.

Participants:

This pilot randomized controlled trial will enroll 60 adult patients (aged ≥18 years) undergoing open-heart surgery at St. Paul's Hospital in Vancouver, Canada. Each arm will include 30 patients. Participants must have at least one risk factor for delirium, including being aged 64 or older, a history of delirium, stroke or TIA, cognitive impairment, or depression. Individuals with severe pre-existing cognitive impairments will be excluded.

Intervention:

Participants will be randomized 1:1 to either the Mindful Garden intervention or standard care. Due to the nature of the intervention, blinding is not feasible. In the intervention group, the Mindful Garden device will be made available for up to 7 days postoperatively or until discharge. All participants will receive standard post-operative care, including routine non-drug delirium prevention measures.

Outcomes:

Primary feasibility outcomes include recruitment success, adherence to study protocol, and participant satisfaction. Secondary clinical outcomes involve:

* Frequency of unscheduled psychotropic medication use
* Incidence and severity of delirium (measured via the Intensive Care Delirium Screening Checklist and Confusion Assessment Method)
* Agitation (Richmond Agitation Sedation Scale)
* Anxiety (State Trait Anxiety Inventory)
* Recovery quality (QoR-15 score)
* Presence of Hallucinations (PSYRATS)
* Hospital length of stay

Anticipated Impact:

This pilot trial will assess whether integrating the Mindful Garden device into post-cardiac surgery care is practical and beneficial. Results will inform a larger trial and may support broader implementation of non-pharmacological digital therapeutics to enhance recovery, reduce delirium, and minimize reliance on psychoactive drugs in surgical settings.

ELIGIBILITY:
Inclusion Criteria:

* Planned open-heart cardiac surgery (e.g. coronary artery bypass grafting, valve replacement surgery);
* Able to understand study procedures and provide informed consent in English;
* At least one delirium risk factor: 1) Age less than 65yrs; 2) History of delirium; 3) History of stroke/TIA; 4) Known cognitive impairment; 5) Depression requiring medication.

Exclusion Criteria:

* Severe pre-existing cognitive impairment (Montreal Cognitive Assessment [MOCA6]<10)
* Uncorrected visual impairment;
* Significant impairment from psychiatric disease;
* Enrolment in another clinical trial which may interfere with the study outcome measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Day 0
Adherence to Protocol Rate | Day 30 post surgery
Time Spent with Device | Day 7 post surgery or discharge, whichever comes first
Patient Satisfaction and Perceived Benefits | Day 7 post surgery or discharge, whichever comes first
  Using a Likert Scale in a patient satisfaction questionnaire. The Likert Scale uses 1 as Strongly Disagree and 5 as Strongly Agree.

SECONDARY OUTCOMES:
Incidence and Severity (days) of Delirium | Twice daily until Day 7 post surgery or discharge, whichever comes first
  Measured by the Intensive Care Delirium Screening Checklist in the CSICU and the Confusion Assessment Method after discharge to the ward.
Number of Unscheduled Psychoactive Medications or IV Infusions | Day 7 post surgery or discharge, whichever comes first
  Examples of medications are haloperidol, loxapine, and dexmedetomidine
Agitation in CSICU | Every 4 hours while admitted to CSICU
  Measured using the Richmond Agitation Sedation Scale:
  Positive scores (+1 to +4): Indicate increasing agitation or restlessness. Negative scores (-1 to -5): Indicate increasing levels of sedation or unconsciousness.
  A score of 0: represents the desired state of alertness and calmness
Patient reported outcomes of anxiety | Day 0, 3, 30 post surgery
  Patient reported outcomes of anxiety will be measured using the State Trait Anxiety Inventory. The State Trait Anxiety Inventory consists of 40 items in total. 20 items for State Anxiety (S-Anxiety) range 20-80 and 20 items for Trait Anxiety (T-Anxiety) range 20-80.
Length of CSICU and hospital stays (days) | Day 30 or day of discharge, whichever comes first
Patient reported Quality of Recovery | Day 0, 3, 30 post surgery
  Measured using Quality of Recovery (QoR-15). Patients score items on a 1 to 5 scale with 1 being Not at All and 5 being Extremely. These scores are totalled where 15-30 indicates Poor Quality of Recovery, 31-50 indicates Moderate Quality of Recovery, and 51-75 indicates Good Quality of Recovery.
Presence of hallucinations and delusions | Day 3 post surgery
  Measured using the Psychotic Symptom Rating Scales (PSYRATS). PSYRATS has 2 subscales: Auditory Hallucinations (AH) and Delusions (D). AH has 11 items each scored 0-4 with a sum of 0 indicating no symptoms and a sum of 44 indicating most severe symptoms. D has 6 items each scored 0-4 with a sum of 0 indicating no symptoms and a sum of 24 indicating most severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Alana Flexman, MD MBA, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Confidentiality restrictions from institution.

REFERENCES:
- [Background] Nicholas M, Wittmann J, Norena M, Ornowska M, Reynolds S. A randomized, clinical trial investigating the use of a digital intervention to reduce delirium-associated agitation. NPJ Digit Med. 2023 Oct 30;6(1):202. doi: 10.1038/s41746-023-00950-4. PMID 37903857
- [Background] Tse L, Schwarz SK, Bowering JB, Moore RL, Barr AM. Incidence of and Risk Factors for Delirium After Cardiac Surgery at a Quaternary Care Center: A Retrospective Cohort Study. J Cardiothorac Vasc Anesth. 2015 Dec;29(6):1472-9. doi: 10.1053/j.jvca.2015.06.018. Epub 2015 Jun 12. PMID 26395395